CLINICAL TRIAL: NCT05169086
Title: The Effectiveness of the Elastic Component of the Multilayer Bandage in the Treatment of Patients With Lymphedema at the University Hospital of Montpellier : a Randomised Clinical Study
Brief Title: Comparison of Two Types of Bandages in the Treatment of Lymphoedema
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0620
Record Dates: First submitted 2021-11-17; First posted 2021-12-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Lymphoedema
Keywords: Lymphology; Chronic disease; reduction bandages
MeSH Terms: conditions — Lymphedema; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a cohort study of patients at the University Hospital during the first two days of intensive treatment. The patients are randomly divided into two groups (N=10).

Throughout the study, group A is treated with the multilayer elastic bandage while group B is bandaged with contention only. The bandages were applied on the first and second day and were maintained in place. The bandages were applied on the first and second day and were maintained for 24 hours. All patients performed 30 minutes of physical activity in the bandage on both days.

The evaluation is based on the volumetric difference, skin quality and quality of life of these patients

ELIGIBILITY:
Inclusion criteria:

* Adult with unilateral lower limb lymphoedema
* Stage 2 or 3 lymphoedema
* 1st intensive decongestant treatment
* Ability to sit on a cycloergometer

Exclusion criteria:

* Severe cardiac disease
* Infectious dermoepidermitis
* Bandage unbearable for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients with primary or secondary lymphedema receiving intensive decongestant treatment at the Montpellier University Hospital. Patients must be of legal age and have unilateral stage 2 or 3 lymphedema.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Perimetry of the affected limb | day 1
  The physiotherapist measures the perimeter of the limb with a tape measure
Perimetry of the affected limb | Day 2
  The physiotherapist measures the perimeter of the limb with a tape measure
Volumetry of the affected limb | day 1
  the volume is calculated using computer software.
Volumetry of the affected limb | Day 2
  the volume is calculated using computer software.

SECONDARY OUTCOMES:
Quality of life questionnaire | day 1
  The patient completes the Lymphoedema Quality of Life Questionnaire (LYMQUOL leg) on admission to the ward and by email one month later
Quality of life questionnaire | one month later
  The patient completes the Lymphoedema Quality of Life Questionnaire (LYMQUOL leg) on admission to the ward and by email one month later

CONTACTS AND LOCATIONS:
Overall Officials: nicolas Erdocio, student, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC